CLINICAL TRIAL: NCT00954759
Title: The Effect of Chiropractic Treatment on Infantile Colic A Randomized, Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Abandoned due to poor recruitment
Sponsor: Nordic Institute of Chiropractic and Clinical Biomechanics (Other)
Collaborators: Foundation for the Advancement of Chiropractic Research (Unknown); University of Southern Denmark (Other)
Responsible Party: Lise Hestbaek, senior researcher, Nordic Institute of Chiropractic and Clinical Biomechanics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCT Colic; CVK S-20090056
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Infantile Colic
Keywords: Infantile colic; Chiropractic; Manipulation; Randomized controlled trial
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chiropractic treatment (Experimental): Manipulation and/or mobilisation
  Interventions: Procedure: Chiropractic treatment
- Visit without active treatment (Placebo Comparator): The child is brought in for chiropractic treatment, but no active treatment is delivered. The parents are unaware whether treatment is delivered or not.
  Interventions: Procedure: Visit without active treatment

INTERVENTIONS:
Procedure: Chiropractic treatment
  Other Names: Manipulation, mobilisation
  Arms: Chiropractic treatment
Procedure: Visit without active treatment — The child is brought in for chiropractic treatment, but no active treatment is delivered. The parents are unaware whether treatment is delivered or not.
  Arms: Visit without active treatment

SUMMARY:
Infantile colic is a condition that affects more than 10% of babies and their families. The reason, and hence the proper treatment, for this condition is unknown and many causes have been suggested. One of the treatments that parents choose is chiropractic manipulation. In Denmark, around 4,000 babies are treated for colic by chiropractors each year although the effect of chiropractic treatment of infantile colic has not been properly scientifically evaluated.

The effect of chiropractic treatment on infantile colic needs to be investigated since this is a very common disorder with no known effective treatment but with good empirical evidence of the value of chiropractic treatment. Although it is usually considered to be a benign and self-limiting condition, some studies suggest there might be long-term effects in terms of psychomotor problems. In worst case, the infants' crying may also lead to violence and 'shaken baby syndrome'.

Null hypothesis: There is no effect of chiropractic treatment on the course of infantile colic.

This study is a controlled clinical trial, where infants fulfilling the diagnostic criteria for colic will be randomized into two groups. One group will receive treatment and the other won't. This will determine the overall effect and furthermore, subgroup analyses will be performed to identify possible subgroups of infants who will benefit the most from the treatment.

The results from subgroup analyses can help to identify children who might benefit from the treatment. Then treatment can be initiated early and a lot of hardship can be avoided for both the babies and the families.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary: To investigate the effect of chiropractic treatment on infantile colic.

Secondary: A) To investigate if infants with suspected musculoskeletal problems respond differently to the treatment than those without. B) To investigate whether health visitors and chiropractors can agree on the diagnosis of "suspected musculoskeletal problems".

METHOD:

A randomized controlled single blind multicenter clinical trial with a nested case-crossover study.

Infants fulfilling the diagnostic criteria for colic will be recruited by health visitors and randomized to chiropractic treatment or no treatment. The parents will be unaware of the child's allocation. All children will be taken to the chiropractors' treatment room while the parents stay in the reception areas. Before treatment, both the recruiting health visitors and the chiropractors will note, whether they suspect musculoskeletal involvement or not. All analyses will be adjusted for known confounders, which will be recorded by the health visitor at baseline.

PERSPECTIVE FOR HEALTH CARE:

First of all, the study will evaluate the effect of chiropractic treatment of infantile colic. Secondly, it will clarify if the treatment effect differ between children with suspected musculoskeletal problems and those without. If children with musculoskeletal problems respond better to chiropractic treatment than others, the study will also indicate whether the health nurse is able to identify these children.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-10 weeks.
* Minimum crying and fussing: three hours per day, three days per week.

Exclusion criteria:

* Known disease.
* Unsatisfying weight gain.
* Psychological or developmental compromise.
* Contraindications for chiropractic treatment.

Ages: 2 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Decrease in hours of crying | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lise Hestbaek, PhD, Study Director — Nordic Institute of Chiropractic and Clinical Biomechanics
Locations (1):
- Nordic Institute of Chiropractic and Clinical Biomechanics, Odense, DK, Denmark